CLINICAL TRIAL: NCT06197581
Title: Safety Assessment of Concurrent Radiotherapy and Novel Systemic Therapy for Breast Cancer
Acronym: RADIOCOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yirui Zhai,MD., Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4214；Approve No.23/384-4216
Record Dates: First submitted 2023-12-05; First posted 2024-01-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer, Familial Male; Radiotherapy; Complications; Chemotherapeutic Toxicity; Immune Checkpoint Inhibitor; CDK4/6 Inhibitor; Trastuzumab; Pertuzumab; PARP Inhibitor
Keywords: Breast Cancer; Radiotherapy; Adverse events; Capecitabine; Trastuzumab; Pertuzumab; Immune checkpoint inhibitor; CDK4/6 inhibitor; PARP inhibitor
MeSH Terms: conditions — Breast Cancer, Familial Male; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RT+capecitabine (Other): Patients will receive concurrent radiotherapy and capecitabine.
  Interventions: Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients)
- RT+HER2 inhibitors (Other): Patients will receive concurrent radiotherapy and any HER2 inhibitors ( eg. trastuzumab plus pertuzumab or TDM1)
  Interventions: Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients)
- RT+ CDK4/6 inhibitors (Other): Patients will receive concurrent radiotherapy and any of the CDK4/6 inhibitors (abemaciclib，palbociclib ,ribociclib or other CDK4/6 inhibitors)
  Interventions: Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients)
- RT+PARP inhibitor. (Other): Patients will receive concurrent radiotherapy and PARP inhibitor(Olaparib or other PARP inhibitors)
  Interventions: Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients)
- RT+ICI (Other): Patients will receive concurrent radiotherapy and immune checkpoint inhibitor (Pembrolizumab or other anti-PD1/PDL1 regimens).
  Interventions: Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients)

INTERVENTIONS:
Radiation: Chest wall / breast radiation with or without lymph node region radiation.(For all of the enrolled patients) — Patients will receive chest wall / breast radiation with or without lymph node region radiation and novel drugs(for specific population according to guidelines) concurrently.
  Other Names: capecitabine（For Arm RT+capecitabine）; HER2 inhibitors (For Arm RT+HER2 inhibitors); CDK4/6 inhibitors(For Arm RT+CDK4/6 inhibitors); PARP inhibitors（For Arm RT+PARP inhibitor）; ICIs(For RT+ICI)

SUMMARY:
Radiation therapy is a crucial part in the comprehensive treatment of breast cancer. In recent years, emerging systemic treatment regimens such as HER 2 inhibitors, CDK 4/6 inhibitors, PARP inhibitors, capecitabine and PD1 inhibitors have greatly improved the prognosis of breast cancer and has become the standard treatment for specific populations. A considerable number of patients require both radiotherapy and maintenance systemic therapy. However, it is not clear whether systemic therapy should be synchronized or suspended in radiotherapy，despite that previous basic research shows that some molecular drug therapy and radiotherapy has a clear synergy mechanism. There is an agent need for a definite evidence to evaluate the safety of synchronous treatment, to support clinical diagnosis and treatment and the next step of comprehensive treatment. The implementation of the new radiotherapy technology represented by IMRT takes into account the prescription dose homogenization and the minimization of normal tissue dosage, which provides a certain basis for the combination therapy. Based on the above conditions, this study intends to enroll patients between 18 and 70 years old with chest wall / breast ± lymphatic drainage area and requiring capecitabine, CDK 4/ 6 inhibitor, HER2 targeted therapy or immunotherapy. Radiation and novel systemic therapies would be delivered concurrently. The study aimed at evaluating the safety of combined treatments.

ELIGIBILITY:
Inclusion Criteria:

ECOG 0-2. Aged 18-70 years old. Pathologically diagnosed as breast cancer. Need to receive radiotherapy according to guidelines. Radiotherapy target volume included chest wall/breast with or without lymph node regions.

Need to receive one of the following therapies according to guidelines, capetabine, CDK4/6 inhibitor, PARP inhibitor , ICIs , HER2 inhibitors.

Exclusion Criteria:

Male breast cancer. Allergy to the upper medicines before. Will receive trastuzumab alone during and/or after radiotherapy. With severe other disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Grade 3 adverse events | Every week during the radiation , week 4 and week 12 after radiation, and at any time when severe symptoms were recorded within 3 months after radiation.
  To investigate the adverse events and safety of the combined treatment.

SECONDARY OUTCOMES:
Adverse events with any grade | Every week during the radiation , week 4 and week 12 after radiation, and at any time when severe symptoms were recorded within 3 months after radiation
  To investigate the adverse events and safety of the combined treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yirui Zhai, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Bo Lan, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shulian Wang, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Fei Ma, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital ,National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Minckwitz G, Procter M, de Azambuja E, Zardavas D, Benyunes M, Viale G, Suter T, Arahmani A, Rouchet N, Clark E, Knott A, Lang I, Levy C, Yardley DA, Bines J, Gelber RD, Piccart M, Baselga J; APHINITY Steering Committee and Investigators. Adjuvant Pertuzumab and Trastuzumab in Early HER2-Positive Breast Cancer. N Engl J Med. 2017 Jul 13;377(2):122-131. doi: 10.1056/NEJMoa1703643. Epub 2017 Jun 5. PMID 28581356
- [Result] Tutt ANJ, Garber JE, Kaufman B, Viale G, Fumagalli D, Rastogi P, Gelber RD, de Azambuja E, Fielding A, Balmana J, Domchek SM, Gelmon KA, Hollingsworth SJ, Korde LA, Linderholm B, Bandos H, Senkus E, Suga JM, Shao Z, Pippas AW, Nowecki Z, Huzarski T, Ganz PA, Lucas PC, Baker N, Loibl S, McConnell R, Piccart M, Schmutzler R, Steger GG, Costantino JP, Arahmani A, Wolmark N, McFadden E, Karantza V, Lakhani SR, Yothers G, Campbell C, Geyer CE Jr; OlympiA Clinical Trial Steering Committee and Investigators. Adjuvant Olaparib for Patients with BRCA1- or BRCA2-Mutated Breast Cancer. N Engl J Med. 2021 Jun 24;384(25):2394-2405. doi: 10.1056/NEJMoa2105215. Epub 2021 Jun 3. PMID 34081848
- [Result] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Result] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola A, Tanner M, Ahlgren J, Auvinen P, Lahdenpera O, Villman K, Nyandoto P, Nilsson G, Poikonen-Saksela P, Kataja V, Bono P, Junnila J, Lindman H. Adjuvant Capecitabine for Early Breast Cancer: 15-Year Overall Survival Results From a Randomized Trial. J Clin Oncol. 2022 Apr 1;40(10):1051-1058. doi: 10.1200/JCO.21.02054. Epub 2022 Jan 12. PMID 35020465